CLINICAL TRIAL: NCT02688998
Title: Simple, Prospective and Randomized Trial to Obtain Answers to Questions of Standard of Care: Vascular Access Strategies for (Neo) Adjuvant Breast Cancer Treatment Without Trastuzumab: A Study From the REthinking Clinical Trials Program (REaCT-vascular Access Her2 Negative).
Brief Title: REaCT-vascular Access Her2 Negative Vascular Access Strategies for (Neo) Adjuvant Breast Cancer Treatment Without Trastuzumab
Acronym: OTT 15-07
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20160006-01H
Record Dates: First submitted 2016-02-18; First posted 2016-02-23 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer; Cancer
Keywords: HER2 negative
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Catheterization, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Venous access PORT or PICC (Active Comparator): Participants will receive a central line placement either a PORT or a PICC prior to the initiation of chemotherapy.
  Interventions: Device: venous access PORT or PICC
- No intervention (No Intervention): Participants will only receive a central line if required once chemotherapy has been initiated.

INTERVENTIONS:
Device: venous access PORT or PICC — Participants will receive a venous access prior to starting chemotherapy
  Arms: Venous access PORT or PICC

SUMMARY:
In the REaCT-Vascular Access Her2 negative study, the investigator will use a novel method to allow comparisons of established standard of care vascular access strategies using the "integrated consent model" as part of a pragmatic clinical trial.

Determining the optimal vascular access strategy remains an important medical issue for patients, nurses, physicians and society. A novel method to allow comparison of established standards of care is needed as part of an increasing internationally mandated incentive to perform more pragmatic clinic trials.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary breast cancer
* Planned to start either FEC-D, AC-D, dose-dense AC-T, TAC, or TC chemotherapy, in the adjuvant or neoadjuvant setting.
* ≥19 years of age
* Able to provide verbal consent

Exclusion Criteria:

• Contraindication to central line placement.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-04; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Accrual rates | One year
  Percentage of patients who receive (neo)adjuvant IV systemic therapy for Her 2 negative breast cancer compared to the number of participants who agree to randomization. The total number of new patients receiving (neo) adjuvant IV systemic cytotoxic therapy will be provided by the local chemotherapy pharmacy and Oncology Patient Information System records.
Patient compliance | One year
  Percentage of participants who are randomized who accept randomization, and percentage of patients who cross-over to receive a central line while on study will be calculated using the chemotherapy treatment documentation in the designated hospital electronic patient record program

SECONDARY OUTCOMES:
Physician engagement | One year
  Percentage of medical oncologists who have agreed to participate in the trial compared to the percentage who approached patients regarding the trial.
Rates of thrombotic events | One year
  2. Rates of documented thrombotic events need for anticoagulation, line infections, phlebitis, and extravasations during chemotherapy.
Number of attempts at cannulation | One year
  3. For those patients randomised to peripheral access information on the number of attempts at cannulation will be collected and site of cannulation. (ipsilateral to surgery vs contralateral to surgery)

CONTACTS AND LOCATIONS:
Locations (1):
- The Ottawa Hospital Cancer Centre, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Robinson A, Stober C, Fergusson D, Kehoe A, Bedard D, MacDonald F, Brunet MC, Saunders D, Mazzarello S, Vandermeer L, Joy AA, Awan A, Basulaiman B, Mallick R, Hutton B, Clemons M; REaCT investigators. A multicentre, randomized pilot trial comparing vascular access strategies for early stage breast cancer patients receiving non-trastuzumab containing chemotherapy. Breast Cancer Res Treat. 2019 Nov;178(2):337-345. doi: 10.1007/s10549-019-05388-5. Epub 2019 Aug 7. PMID 31392518